CLINICAL TRIAL: NCT04209036
Title: 2D Versus 3D Total Laparoscopic Hysterectomy by Surgeons in Training: a Prospective Randomized Trial
Brief Title: Can 3D Laparoscopy Improve Surgical Performances in Surgeons in Training?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Other Study IDs: CICOG-30-10-19\48
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Uterine Fibroid; Uterine Bleeding; Uterine Prolapse
Keywords: 3D laparoscopy; 2D laparoscopy; surgeons in training
MeSH Terms: conditions — Leiomyoma; Uterine Hemorrhage; Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D laparoscopy arm: patients submitted to total hysterectomy using a 3D laparoscopic camera
  Interventions: Other: 0° 3D laparoscopy high-definition camera(Olympus Winter & IBE GMBH, Hamburg - Germany)
- 2D laparoscopy arm: patients submitted to total hysterectomy using a 2D laparoscopic camera (standard laparoscopic camera)

INTERVENTIONS:
Other: 0° 3D laparoscopy high-definition camera(Olympus Winter & IBE GMBH, Hamburg - Germany) — total laparoscopic hysterectomy using a 3D laparoscopy high-definition system
  Groups: 3D laparoscopy arm

SUMMARY:
Due to the inconclusive results on the benefits of 3D laparoscopic system present in literature, this prospective randomised pilot study aims to assess if the operative time of total laparoscopic hysterectomy (TLH) for benign indication performed by trainees could be reduced using 3D laparoscopy instead of standard laparoscopy.

DETAILED DESCRIPTION:
All patients with benign uterine pathology at preoperative examinations (pelvic ultrasound and/or magnetic resonance and/or CT scan) and with indication for total laparoscopic hysterectomy, will be enrolled in the study.

While under general anesthesia, the patient is positioned in the dorsal lithotomic position with both legs supported in stirrups with a Trendelenburg tilt and arms along the body. A four disposable or reusable, sterile trocar transperitoneal approach is used. A 10 mm port is inserted at the umbilicus for the telescope. Once pneumoperitoneum (12 mmHg) is achieved, intra-abdominal visualization will be obtained with a 0° high-definition telescope (HD EndoEye 10 mm, Olympus Winter & IBE GMBH, Hamburg - Germany) or with 0° 3D laparoscopy high-definition (Olympus Winter & IBE GMBH, Hamburg - Germany). The instruments used include bipolar grasper, monopolar scissors, monopolar hook, various graspers and a suction irrigation system. Clermont Ferrand uterine manipulator (Model K.Storz Endoskope,Tuttlingen, Germany) is optionally used to move the uterus.

Total hysterectomy is then performed according to standard technique used by the recruiting center (development of the pararectal space and identification of uterine artery, coagulation of ovarian pedicles, development of the vesico-uterine septum, colpotomy).The vaginal vault is then closed with a 0 Vycril suture laparoscopically (continuous suture).

Detailed operative time, intra and post operative early complications will be recorded (Extended Clavien-Dindo classification of surgical complications will be used for post operative complications)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from benign uterine pathology (uterine fibromatosis, abnormal blood loss, complex hyperplasia with atypia, uterine prolapse) with indication for total uterine hysterectomy
* Uterine size </= than 15 cm
* American Society of Anesthesiologists (ASA) class < 3
* Patient's informed consent
* No actual pregnancies or pelvic inflammatory disease
* No previous major abdominal surgical procedures

Exclusion Criteria:

* Suspected neoplastic pathology
* Patients not eligible for surgery

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: All patients with benign uterine pathology at preoperative examinations (pelvic ultrasound and / or magnetic resonance and / or abdominal CT scan) and with indication for total laparoscopic hysterectomy, will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | intra-operative
  To compare operative time for Total Laparoscopic Hysterectomy with 3D laparoscopy vs. conventional laparoscopy

SECONDARY OUTCOMES:
Intra-operative complications | intra-operative
  • Evaluate the incidence of intraoperative complications in the two laparoscopic system (intraoperative blood loss, need for intraoperative transfusions, bladder lesions, ureteral lesions, vascular lesions, intestinal lesions)
Early post-operative complications | from surgery up to 30 days from surgery
  Evaluate the incidence of postoperative complications (need for postoperative transfusions, dehiscence of the vaginal cuff, fever, urinary tract infections, surgical wound infections)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fanfani, Professor, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Restaino S, Vargiu V, Rosati A, Bruno M, Dinoi G, Cola E, Moroni R, Scambia G, Fanfani F. 4K versus 3D total laparoscopic hysterectomy by resident in training: a prospective randomised trial. Facts Views Vis Obgyn. 2021 Sep;13(3):221-229. doi: 10.52054/FVVO.13.3.027. PMID 34555876